CLINICAL TRIAL: NCT00787748
Title: COPD and Cardiovascular Risk in the Population
Acronym: CORSAIB
Status: Completed | Type: Observational
Sponsor: Cimera (Network)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Other Study IDs: PI061228; IB-9949; IB-615/06PI
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Cardiovascular Disease
Keywords: Cardiovascular; COPD; Population; Prevalence; Underdiagnosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Samples of serum were frozen at -80 ºC
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The prevalence of chronic obstructive pulmonary disease (COPD) in patients with cardiovascular disease (CVD) is unknown, and whether or not COPD is adequately diagnosed and treated in these patients has not been investigated before.

We hypothesized that the prevalence of COPD would be significantly higher (30%) in patients with CVD than in the general population. Besides, we anticipated that COPD, a potentially treatable CV risk factor, would be undiagnosed in more than 80% of CVD patients.

DETAILED DESCRIPTION:
We aim to compare clinical and spirometric data in three groups of individuals. Two of them are participants in an ongoing population-based study (CORSAIB) aimed at investigating the distribution of CVD risk factors in the general population of the Balearic Islands, Spain. The design and full methodological details of the CORSAIB study have been published elsewhere (Rigo F, et al. Rev Clin Espa 2005). A third group will include patients with stable CVD regularly visited at the referral hospital of our community.

Inclusion criteria for the study are male and female individuals, aged 40 to 81 years, residents of the Balearic Islands, and who are willing to participate in this research.

ELIGIBILITY:
Inclusion Criteria:

* residents of the Balearic Islands
* willing to participate in this research
* able to sign the written consent form

Exclusion Criteria:

* none

Ages: 40 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Random population sample, and a sample of hospital cardiovascular patients
Sampling Method: Probability Sample
Enrollment: 623 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of COPD defined according to the current GOLD guidelines as a post-bronchodilator forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) <0.7. | Current

SECONDARY OUTCOMES:
Underdiagnosis of COPD | Current
Undertreatment of COPD | Current

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rigo, MD, Study Director — Atención Primaria de Mallorca; Alvar Agusti, MD, Study Director — Cimera
Locations (1):
- CIMERA, Bunola, Balearic Islands, Spain

REFERENCES:
- [Result] Soriano JB, Rigo F, Guerrero D, Yanez A, Forteza JF, Frontera G, Togores B, Agusti A. High prevalence of undiagnosed airflow limitation in patients with cardiovascular disease. Chest. 2010 Feb;137(2):333-40. doi: 10.1378/chest.09-1264. Epub 2009 Sep 25. PMID 19783666